CLINICAL TRIAL: NCT02287155
Title: Occupation Based Health-Promotion Program for People Aged Over 60: "Bliib Gsund"
Acronym: bg60
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Julie Page (Other)
Collaborators: Occupational therapy practice ergoalltag (Unknown); Linthpraxen GmbH (Unknown); Stiftung für Ergotherapie Zürich (Unknown); ErgotherapeutInnen Verband Schweiz evs (Unknown)
Responsible Party: Sponsor-Investigator, Julie Page, Prof., Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZHAW-F&E-Ergo
Record Dates: First submitted 2014-10-16; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: Health Promotion; Intervention Study; Occupational Therapy; Rural Population; Quality of life; Sense of coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- occupation based health promotion (Experimental): The description of the health promotion intervention is provided in the "detailed description" of the study. It's a single arm study.
  Interventions: Behavioral: occupation based health promotion

INTERVENTIONS:
Behavioral: occupation based health promotion — The description of the intervention is provided in the "detailed description" of the study.

SUMMARY:
As in many other countries in the world, the population in Switzerland is growing older. This also means an expansion of costs in the health system. Therefore, the investigators need to find concepts of health promotion to prevent people from getting ill and dependent of the health care system.

Our project aims at developing a health promotion program for persons over 50 years of age in a rural area of Switzerland. The program's name is "bliib gsund". This occupational-therapy directed health promotion program is conducted over a period of six months in two groups of eight persons each. The aim of the program is to enhance the quality of life of the participants, to mediate the competence of integrating health-promoting aspects in their daily life, and to maintain their independence in their life as long as possible. Persons over 50 often find themselves in a phase of transition in life, such as starting retirement, the loss of family members or children moving out. This program will provide them with the ability to continue their lifestyle in a more active way. It embraces topics such as more active pursuits of interests and carrying out personally meaningful activities.

In preparation of the program, the investigators conducted a needs analysis to identify the needs relating to health-promoting offers of the inhabitants living in the specified region. The results showed a high interest and need for such programs. They also helped us to identify several relevant issues to be included in the presented health-promotion program: physical exercise in daily life, healthy nutrition, getting acquainted with new technologies, fall-prevention training and maintaining social contacts. The researchers and the designated occupational therapist, who will be the moderator of the program, can develop the program based on these results.

The evaluation of the program should identify the effect of the program concerning the promotion of self-efficacy, the sense of coherence, quality of life and the program objectives. A questionnaire will be distributed before the program, immediately after and six months after the program.

DETAILED DESCRIPTION:
1. Background

   In Switzerland, the proportion of over-fifty-year-olds is growing rapidly - between 1996 and 2007, the proportion of people over 50 in employment grew from 26% to 31%. By 2020, the proportion will increase to one-third (Meyer, 2008). In addition, the baby boomers will retire in the next few years. In the canton of Glarus, about 26% will be older than 65 years in 2030, compared to only 18% today. The use of health services and the consequential higher costs for the health system will rise dramatically (Cruz et al., 2014). It is believed that approximately 2 billion Swiss Francs could be saved by 2030 by means of health promotion and disease prevention programs in this age group (Stuck et al., 2009). In 2007, the Federal Council designed the "Strategies for the Swiss old-age policy", which is based on the assumptions of "active aging" by the WHO in 2002. The knowledge gained showed that in particular individual health literacy and behavioral and relationship-oriented health promotion efforts strengthen the health and social integration. Moreover, the Federal Council describes that health promotion and the prevention of chronic diseases and functional disability will be future needs (Rielle, Wirz, & Wiesli, 2010). This is supported by the data available from the Federal Office of Statistics, which identified a permanent health problem by 43.2% among 55-64 year olds and 47.2% among 65-74 year olds (BFS, 2012).

   For the above mentioned reasons the existing LINTHPRAXEN Medical Center is expanding their facilities and services in the form of a prevention center. One part of the expansion is creating an occupational therapy-led health promotion program. The program is based on the essential components of the already existing programs "Tatkraft - Gesund im Alter durch Betätigung" (Ferber et al., 2012) "Lifestyle Matters" (Mountain et al., 2008) and "Life-Redesign-Prgram" (Jackson et al., 1998, Hay et al., 2002, Clark et al., 2012) .

   A demand for this program can be seen especially in the municipality of Glarus Süd. According to the "Report on the aging policy in the cantons" of Rielle et al. (2010) the Canton of Glarus and the municipality of Glarus Süd carry out a barely effective age policy. The report lists the relevant issues as: living in old age, health / prevention, finances, volunteer work, social integration and the maintaining of independence of the elderly. When implementing an age strategy, the community setting is of great importance. The "Model Health Canton Glarus", published in February 2014, reflects the problematic situation of the aging population in Glarus and defines principles that describe strategies for health care. Among other things, the Canton aims to expand the health promotion and prevention services and to link local players in health care (Cruz et al. 2014). The project "bliib gsund" is therefore a suitable first initiative in this area.
2. Program objectives

   The program objectives are primarily aimed at learning skills to integrate health-promoting aspects in daily life and to maintain the quality of life (strengthen the sense of coherence, increase quality of life, increase self-efficacy). The main aspect is to maintain the autonomy and independence of the people in everyday life as long as possible.
3. Intended Curriculum

   The main aspect of this study is the pilot implementation of the health-promoting program "bliib gsund". The approach chosen is based on participation to increase the chances of the program to be based on the specific needs of the target audience and to be able to recruit enough participants (at least five to eight) and to communicate the program content effectively. Paying close attention to the needs of the participants concerning program development via a needs analysis increases the chances of success. The project steps are thus as described below.

   3.1 Needs Analysis

   For the needs analysis, existing patients (older than 50) of the LINTHPRAXEN Medical Center health center were interviewed about their expectations of and interests in health-promoting services. The aim was to identify how and by what measures the participants feel best addressed. The questions' structure was mostly nominal scales and semi-open to give the respondents the opportunity to state their individual response (Porst, 2011).

   We sent 2'000 questionnaires to 1'000 households, of which 265 (13.3%) were sent back and then evaluated. This response rate is considered satisfying. Of the 265 responding persons, 162 are women and 93 men. The age distribution shows that 147 persons are aged 50-64, 105 between 65-79 years and four persons are over 80 years of age.

   The questions that dealt with the "bliib gsund" program showed that 43.4% were interested in taking part in it. The reasons for not being interested were participation in other activities or lack of time. Topics for the program content specified in the questionnaires were: adequate exercise in everyday life, healthy diet, memory training, getting acquainted with new technologies, skill training, social relationships, getting to know other health promotion programs in the community as well as safety indoors and outdoors. These specifications provide a good program content basis. The financing of the program participation is accepted by the participants. 89.1% would be willing to pay money for such a program. 66.8% would pay 11-20 Swiss Francs per lesson, 22.8% up to 10 Swiss Francs. A subscription of 300 Swiss Francs for the six-month program as well as other options at the LINTHPRAXEN prevention center would be acquired by 64.2% of the people. Of those who are interested in the program, 86.5% would even be willing to acquire the subscription. A large proportion of the potential participants could imagine participating in the program once per week (47.2%), 23.6% once every two weeks and 13.7% one to two times a week.

   These results clearly show that a need exists in the community Glarus Süd. The inhabitants would even be willing to finance the cost of the program and they would make time for it. There were participants from the age groups of 50-64 year olds as well as 65-79 year olds. If as many participants as the survey suggests could actually be recruited for the program (approx. 100 people), they could be split up into groups according to interests and availability during the week. The survey among the potential participants has acquainted them with the program so that recruiting and advertising should be easier. The results of the survey can therefore clearly be rated as very positive and helpful.

   3.2 Program development

   The results of the above described needs analysis are used for the design of the program. Contents and interventions are matched with findings from previous implementation of the program in other countries. The overall planning is carried out by the Zurich University of Applied Sciences (ZHAW) in collaboration with Angelika Beck, an occupational therapist in the region. She also will lead the implementation of the program.

   3.3 Recruitment of program participants

   Potential participants are recruited from the address file of the LINTHPRAXEN Medical Center, through local cooperation partners (Pro Senectute, and occupational therapy practice "ergoalltag", through doctors and public media, i.e. newspapers, posters and flyers). Another access might be through the church and other seniors' organizations. The aim is to reach a group size of up to ten participants. The program might also run parallel courses, separated according to their activity level and program contents.
4. Intended project steps and duration of the project

The time frame of the entire project is set for November 2013 to September 2015. The planning and conceptual design of the study has been processed since November 2013. The actual start of the program is scheduled for January 2015, and it will then run six months with ten participants (per group). The realization of the project will take place in the existing and newly built facilities of LINTHPRAXEN in Linthal. The project phases as follows:

1. Develop project idea (November 2013 to December 2013)

   1. Getting familiar with the project idea, first literature search
   2. Exchange with developers of the program in foreign countries (Germany, Austria, Great Britain, The Netherlands)
   3. Project concept design handed over to Dr. Fasol, including preliminary budget
   4. Meetings / consultation with the client (Dr. Fasol)
2. Needs analysis (December 2013 to April 2014)

   1. Postal survey (devise questionnaire content and layout, questionnaire distribution)
   2. Systematize results (for further financial requests, for feedback to participants, for feedback to the client)
3. Devise funding applications (December 2013 to March 2014)

   1. Detailed literature search, composing of individual applications
   2. Funding applications
4. Adaption of the program "bliib gsund" for Glarus Süd (May 2014 to November 2014)

   1. Business plan for the offer
   2. Contracting staff / occupational therapist in program
   3. Adapting the content of the program in accordance with needs analysis
   4. Find local cooperating partners (information sheet, establish contact, information meetings for local potential cooperation partners)
   5. Planning evaluation (select survey instruments, adjust evaluation sheets from the German version of the program)
5. Pilot implementation of "bliib gsund" (January 2015 to February 2016)

   1. 12 modules of 90 min; two parallel courses if possible
   2. Ongoing adaptation (preparing for each module)
   3. Evaluation before - after
   4. Evaluation after six months
6. Project completion (January 2016 to March 2016) Transfer program from ZHAW to LINTHPRAXEN
7. Project management (January 2014 to March 2016)

   1. Contracting
   2. Communication (reporting to donors, ZHAW internal communication, local media work, two publications in scientific journals, two conference visits: presentation of the project)

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age
* Healthy or suffering from a mild to moderate disease

Exclusion Criteria:

* Severe dementia
* Severe chronic disease (such as heart disease, metabolic disease, lung disease)
* Immobility (not able to get to the LINTHPRAXEN)
* State after acute illness, injury (e.g. after a recent stroke, myocardial infarction, fractures)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in self efficacy | baseline (before the programm start), after 6 month (end of programm), after 12 month (follow up)
  The participants are asked to fill out the self-efficacy-scale from Schwarzer&Jerusalem (1999).

SECONDARY OUTCOMES:
Change in sence of coherence | baseline (before the programm start), after 6 month (end of programm), after 12 month (follow up)
  The participants are asked to fill out the sence of coherence-scale from Brähler, Schumacher&Strauss (2002).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Page, Prof. Dr., Principal Investigator — Zurich UAS

REFERENCES:
- [Background] Brähler E, Schumacher J, Strauss B. Diagnostische Verfahren in der Psychotherapie. 2002 Bern: Hogrefe Verlag.
- [Background] Ferber R, Dangl H. Grote A, Kölling D, Marotzki U, Rach M, Schmitt R, Weiß, K. Tatkraft - Gesund im Alter durch Betätigung, Programm zur Gesundheitsförderung. 2002 Idstein.
- [Background] Mountain G, Mozley C, Craig C, Ball L. Occupational Therapy led health promotion for older people: feasability of the Lifestyle Matters Programme. British Journal of Occupational Therapy. 2008 71(10), 406-413.
- [Background] Meyer K. Gesundheit in der Schweiz - Nationaler Gesundheitsbericht 2008. In V. H. Huber (Ed.). Bern: Schweizerisches Gesundheitsobservatorium.
- [Background] Stuck AE, Born S, Meyer K. Umsetzung von Programmen zur Gesundheitsförderung und Prävention im Alter nach dem "Gesundheits-Profil Verfahren". In B. f. Statistik (Ed.), obsan fact sheet. 2009. Neuchâtel: Schweizerisches Gesundheitsobsvervatorium.
- [Background] Rielle Y, Wirz R, Wiesli R. Alterspolitik in den Kantonen. In F. f. Gesundheitspolitik (Ed.). 2010. Bern: Fachstelle für Gesundheitspolitik.
- [Background] Probst R. Fragebogen - Ein Arbeitsbuch (Vol. 3. Auflage). 2011. Wiesbaden.
- [Background] Cruz D, Knoth S, Sommer C. Leitbild Gesundheit Kanton Glarus - Vernehmlassung. In D. F. u. Gesundheit (Ed.), 2014 pp. 1-28. Glarus: Departement Finanzen und Gesundheit.
- [Background] BFS. Schweizerische Gesundheitsbefragung 2012 - Übersicht. Retrieved 13.12.2014, from Bundesamt für Statistik. http://www.bfs.admin.ch/bfs/portal/de/index/news/publikationen.html?publicationID=5352
- [Background] Schwarzer R, Jerusalem M. Skalen zur Erfassung von Lehrer- und Schülermerkmalen. Dokumentation der psychometrischen Verfahren im Rahmen der Wissenschaftlichen Begleitung des Modellversuchs Selbstwirksame Schulen. 2009. Berlin: Freie Universität Berlin.
- [Background] Clark F, Jackson J, Carlson M, Chou CP, Cherry BJ, Jordan-Marsh M, Knight BG, Mandel D, Blanchard J, Granger DA, Wilcox RR, Lai MY, White B, Hay J, Lam C, Marterella A, Azen SP. Effectiveness of a lifestyle intervention in promoting the well-being of independently living older people: results of the Well Elderly 2 Randomised Controlled Trial. J Epidemiol Community Health. 2012 Sep;66(9):782-90. doi: 10.1136/jech.2009.099754. Epub 2011 Jun 2. PMID 21636614
- [Background] Hay J, LaBree L, Luo R, Clark F, Carlson M, Mandel D, Zemke R, Jackson J, Azen SP. Cost-effectiveness of preventive occupational therapy for independent-living older adults. J Am Geriatr Soc. 2002 Aug;50(8):1381-8. doi: 10.1046/j.1532-5415.2002.50359.x. PMID 12164994
- [Background] Jackson J, Carlson M, Mandel D, Zemke R, Clark F. Occupation in lifestyle redesign: the Well Elderly Study Occupational Therapy Program. Am J Occup Ther. 1998 May;52(5):326-36. doi: 10.5014/ajot.52.5.326. PMID 9588257